CLINICAL TRIAL: NCT06582823
Title: Effects of a Health Belief Model-Based Community Educational Program to Increase the Awareness of Atrial Fibrillation Among Older Adults: a Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ryan Kin Ho Hui, Doctor of Nursing Student, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: UW 23-344
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention integrate behavioral modeling to promote knowledge and skill retention and uptake. The content of the education sessions is consistent with the clinical management guidelines published by the E
  Interventions: Other: Health belief model-based community educational program
- Control (Active Comparator): The control group
  Interventions: Other: Control

INTERVENTIONS:
Other: Health belief model-based community educational program — The 5-week intervention includes two weekly 60-minute face-to-face sessions for 8-10 participants, two weekly telephone follow-ups, and a booster session.
  Week 1: Focuses on increasing knowledge about atrial fibrillation (AF), its risks, complications, and treatment benefits. The principal investigator (PI) provides education using interactive methods and colored visuals.
  Week 2: Emphasizes skill building for pulse palpation to detect irregular pulses. Participants learn through demonstrations and practice using a simulated arm.
  Weeks 3-4:Telephone follow-ups monitor adherence to pulse checking and address barriers. Support and advice are provided by the PI.
  Week 5: A booster session reinforces knowledge and skills with scenario-based practice and use of a simulated arm.
  Arms: Intervention
Other: Control — The control group will receive an information leaflet presenting information about AF, health risks and complications associated with AF, common methods to screen for AF, and follow-up actions if positive screening results are suspected.
  Arms: Control

SUMMARY:
The goal of this study is to evaluate the effects of a theory-based community educational program among older adults in the community on atrial fibrillation (AF) knowledge. It will also learn about their competency to detect irregular pulses and compliance to regular pulse check. The main questions it aims to answer are:

Do older adults in the community who received the Health Belief Model-based educational program have higher AF awareness?

Researchers will compare the educational program with the control, who receive an information leaflet about AF to see the effect on improving AF awareness.

Participants will:

Receive a 5-week Health Belief Model-based educational program or receive an information leaflet about AF.

Be reassessed immediately post-intervention and 3 month afterwards. Keep a logbook on their compliance to the advice of regular pulse palpation to detect AF pulse .

ELIGIBILITY:
Inclusion Criteria:

* adults aged 65 or older
* without a confirmed diagnosis of AF

Exclusion Criteria:

* cannot read Chinese
* with cognitive impairment (Abbreviated Mental Test ≤ 6)
* physical limitations in performing pulse palpation

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2023-08-12 (Actual); Primary Completion 2024-11-29 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Atrial Fibrillation Knowledge Scale | From enrollment to the end of study at 3 months
  Atrial Fibrillation Knowledge Scale (AFKS-C, Chinese version) is a validated tool that includes 11 items concerning AF knowledge in general (3 items), symptom recognition (3 items), and treatment (5 items). Respondents can choose 1 of 3 options as an answer to each item. Marks will be given for correct answers and no deduction for incorrect answers, and higher marks indicate a higher AF knowledge level. The content validity index of the AFKS-C was 0.94, and the Kuder-Richardson formula 20 value was 0.60, indicating acceptable psychometric properties.
  Li, P. W. C., Yu, D. S. F., Yan, B. P., Hendriks, J. M., Wong, C. W. Y., & Chan, B. S. (2021). Psychometric Validation of the Chinese Version of the Atrial Fibrillation Knowledge Scale in Chinese Patients With Atrial Fibrillation. The Journal of cardiovascular nursing, 38(1), 92-100. https://doi.org/10.1097/JCN.0000000000000881

SECONDARY OUTCOMES:
Competency in differentiating regular and irregular pulses | From enrollment to the end of study at 3 months
  Competency in differentiating regular and irregular pulses will be evaluated by a simulated arm. Participants will be instructed to perform radial pulse palpation on the simulated arm in order to differentiate regular and irregular pulses. A total of four scenarios, with two regular and two irregular pulses, will be set up and randomly presented to evaluate the competency of participants in differentiating the regularity of pulses.
Compliance to performing self-screening of pulses | From enrollment to the end of treatment at 3 months
  Compliance to performing self-screening of pulses is measured by using a logbook. Participants will be instructed to perform twice-daily radial pulse palpation. The regularity and pulse rate will be documented in the logbook. The compliance to the advice of pulse palpation will be evaluated by the frequency of performing pulse palpation and the percentage of completion of the logbook.
Patient Health Questionanire-4 (PHQ-4) | From enrollment to the end of treatment at 3 months
  Patient Health Questionanire-4 (PHQ-4)will be used for measuring anxiety and depression symptoms in the past 14 days. It has 4 items to be rated on a 4-point scale ranging from 0 to 3, with higher sum scores indicating greater psychological distress. The Chinese version of PHQ-4 have good composite reliability (McDonald Omega > 0.8).
  Fong, T. C. T., Ho, R. T. H., & Yip, P. S. F. (2023). Psychometric properties of the Patient Health Questionnaire-4 among Hong Kong young adults in 2021: Associations with meaning in life and suicidal ideation. Frontiers in psychiatry, 14, 1138755. https://doi.org/10.3389/fpsyt.2023.1138755
EuroQol Five Dimensions Five Levels (EQ-5D-5L) | From enrollment to the end of treatment at 3 months
  EuroQol Five Dimensions Five Levels (EQ-5D-5L) will be used to measure health-related quality of life (HRQoL). It consists of two parts: EQ-5D descriptive system and EQ visual analogue scale. The first part uses 5 levels to indicate a participant's health state on 5 dimensions - mobility, self-care, usual activities, pain/discomfort, and anxiety/depression - and the second part is an additional self-rated health item rated on a visual analogue scale ranging from 0-100. The Chinese version of EQ-5D-5L was validated with Cronbach's alpha coefficient 0.78.
  Cheung, P. W. H., Wong, C. K. H., Samartzis, D., Luk, K. D. K., Lam, C. L. K., Cheung, K. M. C., & Cheung, J. P. Y. (2016). Psychometric validation of the EuroQoL 5-Dimension 5-Level (EQ-5D-5L) in Chinese patients with adolescent idiopathic scoliosis. Scoliosis and spinal disorders, 11, 19. https://doi.org/10.1186/s13013-016-0083-x

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Kin Ho HUI, Principal Investigator — School of Nursing, LKS Faculty of Medicine, The University of Hong Kong
Locations (1):
- School of Nursing, LKS Faculty of Medicine, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided